CLINICAL TRIAL: NCT01235039
Title: A Single Center, Double Blind, Randomized Crossover Study Evaluating the Bioequivalence of VIAject®7 Compared to VIAject®25 and Comparing the Pharmacokinetic and Pharmacodynamic Properties of VIAject®7 to Insulin Lispro in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study Evaluating the Bioequivalence of VIAject®7 Compared to VIAject®25 and Comparing the Pharmacokinetic and Pharmacodynamic Properties of VIAject®7 to Insulin Lispro in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VIAject -030J
Record Dates: First submitted 2010-11-02; First posted 2010-11-05 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation A (Experimental): VIAject®25 for subcutaneous application
  Interventions: Drug: VIAject®25
- Formulation B (Experimental): VIAject®7 for subcutaneous application
  Interventions: Drug: VIAject®7
- Formulation C (Experimental): Insulin Lispro for subcutaneous application
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: VIAject®25 — Two vial presentation for reconstitution and single dose of 12 IU subcutaneous injection and 25 IU/mL
  Arms: Formulation A
Drug: VIAject®7 — One vial presentation and single dose of 12 U for subcutaneous injection and 100 IU/mL
  Arms: Formulation B
Drug: Insulin Lispro — One vial presentation and single dose of 12 IU for subcutaneous injection and 100 IU/mL
  Arms: Formulation C

SUMMARY:
The primary objective of this study is to test for bioequivalence of VIAject®7 and VIAject®25 and to compare the pharmacokinetic/Pharmacodynamic/tolerability characteristics of VIAject®7 with those of VIAject®25 and insulin lispro.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥19 to ≤65 years
* Body Mass Index: ≥18 - ≤28 kg/m2
* Diagnosed with Type 1 Diabetes Mellitus for at least 1 year
* Insulin antibody less than or equal to 10 µU/mL at screening
* Non-smoker, defined as no nicotine consumption for at least one year.
* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)

Exclusion Criteria:

* Type 2 Diabetes Mellitus
* C-peptide value of >1.0 ng/mL
* HbA1c value of > 10.0%
* History of hypersensitivity to any of the components in the study medication
* History of severe or multiple allergies
* Treatment with any other investigational drug in the last 3 months before study entry
* Any systemic treatment with drugs known to interfere with glucose metabolism such as systemic corticoids, non-selective beta-blockers, and monoamine oxidase (MAO) inhibitors within 3 months prior to randomization.
* Changes (type of drug or dose) in concomitant medication other than insulin or insulin analogues in the last 3 weeks prior to randomization.
* Use of non-prescription drugs, except routine vitamins, within 3 weeks prior to the first dose of the test drug. Occasional use of paracetamol/acetaminophen is permitted.
* Progressive disease likely to prove fatal (e.g. malignancies)
* Current drug or alcohol abuse, or a history of drug or alcohol abuse which in the opinion of the Investigator will impair subject safety or protocol compliance
* Significant cardiovascular, respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and/or hematological disease as evaluated by the Investigator
* Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with elevated liver enzymes (AST or ALT >2 times the upper limit of normal) or impaired renal function (serum creatinine values above the upper limit of normal) will not be allowed to enter the trial.
* Any serious systemic infectious disease during the four weeks prior to the first dose of study drug, as judged by the Investigator.
* History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose a risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (hemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
* Blood donation within the last 30 days
* A woman who is lactating
* Pregnant women or women intending to become pregnant during the study
* A sexually active woman - not using adequate contraceptive methods (adequate contraceptive measures include: implants, injectables, combined oral contraceptives, hormonal intrauterine device [IUD], sexual abstinence or vasectomized partner)
* Positive serology for HIV, Hepatitis B or Hepatitis C
* Abnormal ECG, safety lab or physical examination results that are deemed clinically significant by the Investigator
* Lack of compliance or other reasons which, in the opinion of the Investigator, prevent the participation of the subject in the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Serum insulin concentration | 0-480 minutes
  Area under the serum insulin concentration curve for the time interval 0-480 min (AUC-INS 0-480) and maximum serum insulin concentration (C-INS max) (VIAject®7and VIAject®25 only)

SECONDARY OUTCOMES:
Serum insulin concentration | 0-240 minutes
  * AUC-INS: area under the serum insulin concentration curve for the time period 0-240 minutes
  * AUC-INS: area under the serum insulin concentration curve for the time period 0 (VIAject® dosing) to the time when the insulin value returns to baseline
Glucose infusion rate | Between 0-240 minutes and 0-480 minutes
  •AUCGIR: area under the glucose infusion rate curve for the following time periods: 0-240, 0-480 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, M.D, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany